| Official Title: | Decision Support for Smoking Cessation in Young Adults With |
|---|---|
| | Severe Mental Illness |
| NCT number: | NCT01779440 |
| <b>Document Type:</b> | Statistical Analysis Plan |
| Date of the | November 24, 2015 |
| Document: | |

We will describe baseline characteristics of the study group. While controlling for any baseline group differences, baseline past 3 months cessation treatment and intention to use treatment, and symptom severity, we will use logistic regression to assess whether EDSS users are more likely to initiate cessation treatment than the users of the control condition. We will calculate the effect size and its confidence interval to plan for a full-scale RCT. Secondary analyses will include similar techniques to assess the differential effect of the interventions on abstinence, as well as theory of planned behavior constructs, including smoking cessation treatment beliefs.